CLINICAL TRIAL: NCT01181570
Title: Efficacy and Safety of Adalimumab in Patients With Psoriasis and Obstructive Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inno-6016; IMM 10-0005 (Other Grant/Funding Number: Abbott (grant))
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Psoriasis; Sleep Apnea, Obstructive
Keywords: psoriasis; adalimumab; obstructive sleep apnea; obesity
MeSH Terms: conditions — Psoriasis; Sleep Apnea, Obstructive; Obesity | interventions — Adalimumab; Mannitol; Citric Acid; Sodium Citrate; 3-lauroyl-glycero-1-phosphate; Sodium Chloride; Polysorbates; Water; Injections; Sodium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab (Experimental)
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab — Patients receive adalimumab 80 mg followed by 40 mg at week 1 and 40 mg every other week (EOW) thereafter.
  Other Names: Humira; mannitol; citric acid monohydrate; sodium citrate; disodium phosphate dihydrate; sodium dihydrogen phosphate dihydrate; sodium chloride; polysorbate 80; water for injection; sodium hydroxide.
  Arms: Adalimumab
Drug: Placebo — Patients will receive 2 injections of placebo at week 0, one injection at week 1 and one injection every other week (EOW) thereafter.
  Other Names: mannitol; citric acid monohydrate; sodium citrate; disodium phosphate dihydrate; sodium dihydrogen phosphate dihydrate; sodium chloride; polysorbate 80; water for injection; sodium hydroxide
  Arms: Placebo

SUMMARY:
This study will evaluate the effect and safety of adalimumab in approximately 20 subjects with mild to moderate psoriasis and sleep apnea and will be conducted in one treatment center located in Montreal.

Patients with psoriasis often have additional disorders such as obesity. Obese patients are more at risk of developing obstructive sleep apnea. This is believed to be caused by both the collapse of upper airways and inflammation (swelling). Adalimumab, a drug currently approved by Health Canada for the treatment of psoriasis, blocks tumor necrosis factor-alpha (TNF-alpha). This chemical is present at higher levels in patients with sleep apnea. It is believed that adalimumab could improve obstructive sleep apnea by lowering the levels of TNF-alpha.

ELIGIBILITY:
Inclusion Criteria:

* Men or women are 18 to 80 years of age at time of consent.
* Has at least a 6-month history of chronic moderate to severe psoriasis and is a candidate for systemic therapy.
* Has a body surface area (BSA) covered with psoriasis of at least 5% or more at Day 0.
* Has a diagnosis of obstructive sleep apnea confirmed by at least 15 episodes/hour of apnea/hypopnea at the polysomnographic testing on Day -2.
* Unless surgically sterile (or at least 1 year post-menopausal), or abstinent, patient (female) is willing to use an effective method of contraception for at least 30 (90 for "c") days before Day 0 and until at least 6 months after the last drug administration. Effective method of contraception are:

  * Condom with spermicidal foam, cream or gel, sponge with spermicidal foam, cream or gel, diaphragm with spermicidal foam, cream or gel
  * Intra uterine device (IUD)
  * Contraceptives (oral or parenteral)
  * Nuvaring
  * Vasectomised partner
  * Same-sex partner
* Negative serum pregnancy test at the screening visit for female patient of childbearing potential only.
* Patient is judged not to have contraindications to adalimumab as determined by the principal investigator based upon the results of medical history, laboratory profile, physical examination and chest X-ray performed at screening.
* Patient will be evaluated for latent tuberculosis (TB) infection with a purified protein derivative (PPD) or a QuantiFERON-TB Gold test and Chest X-Ray (CXR). All patients who previously received TB immunization (BCG vaccination) will have the QuantiFERON-TB Gold test performed. Patient who demonstrates evidence of latent TB infection (either PPD more than or equal to 5 mm of induration or positive QuantiFERON-TB Gold) or suspicious CXR will not be allowed to participate.
* Capable of giving informed consent and the consent must be obtained prior to any study related procedures.
* Patient must be able and willing to self-administer subcutaneous (SC) injections or have a qualified person available to administer SC injections.

Exclusion Criteria:

* Has received medical treatment for sleep apnea in the 6 months preceding Day 0.
* Presence of other skin diseases or skin infections (bacterial, fungal or viral) that may interfere with evaluation of psoriasis or with patient's safety.
* Has a history of an allergic reaction or significant sensitivity to constituents of study drug, including latex (a component of the pre-filled syringe).
* Use of any non-biological systemic therapy for the treatment of psoriasis (including PUVA (psoralen and ultraviolet A)) less than 30 days before Day 0.
* Use of investigational chemical agents within 30 days or five half-lives prior to Day 0, whichever is longer.
* Use of any biological therapy for the treatment of psoriasis less than 90 days before Day 0.
* Current use of oral or injectable corticosteroids or during the study. Inhaled corticosteroids for stable medical conditions are allowed.
* Use of any topical treatments for psoriasis or phototherapy within two weeks prior to Day 0, at the exception of low strength (hydrocortisone and desonide) topical corticosteroid for the face, groin (including genitals) and inframammary areas.
* Has received Anakinra/Kineret within the last 2 weeks prior to Day 0 or is likely to receive Anakinra/Kinaret during the course of the study.
* Has a poorly controlled medical condition, such as uncontrolled diabetes, documented history of recurrent infections, unstable ischemic heart disease, congestive heart failure, recent stroke (within the past 90 days), chronic leg ulcer or any other condition which, in the opinion of the investigator, would put the patient at risk if participating in the study.
* Has a history of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease (e.g. optic neuritis, visual disturbance, gait disorder/ataxia, facial paresis, apraxia).
* Has a history of cancer or lymphoproliferative disease other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
* Has a history of listeriosis, treated or untreated TB, persistent chronic infections, or recent active infections requiring hospitalization or treatment with intravenous anti-infectives within 30 days or oral anti-infectives within 14 days prior to Day 0.
* Has received any live attenuated vaccine 28 days or less before Day 0 or plans to receive one during the study.
* Has hepatitis B or hepatitis C viral infection.
* Has any of the following: hemoglobin ≤ 10 g/L, white blood cell count ≤ 3.0 X 10^9/L, platelet count ≤130 X 10^9/L, ALT ≥ 3 times the upper limit of normal, AST ≥ 3 times the upper normal limit, total bilirubin ≥ 2 times the upper normal limit or creatinine ≥ 150 µmol/L.
* Current use or plan to use anti-retroviral therapy at any time during the study.
* Is known to have immune deficiency or is immunocompromised.
* Current pregnancy or lactation or considering becoming pregnant during the study or for 150 days after the last dose of study medication.
* Has a history of clinically significant drug or alcohol abuse in the last year.
* Is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of sleep apnea per hour. | 56 Days
  Changes from baseline in number of apnea/hypopnea per hour for patients with psoriasis randomized to adalimumab as compared to patients randomized to topical therapy.

SECONDARY OUTCOMES:
Sleep maintenance efficiency | 56 days
  Changes from baseline in sleep maintenance efficiency for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Total wake time | 56 days
  Changes from baseline in total wake time for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo
Percentage of sleep time | 56 days
  Changes from baseline in percentage of sleep time for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Time spent in REM (rapid eye movement) stage. | 56 days
  Changes from baseline in time spent in REM (rapid eye movement) stage for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Time spent in sleep stage N1 | 56 days
  Changes from baseline in time spent in sleep stages N1 for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Time spent in sleep stage N3 | 56 days
  Changes from baseline in time spent in sleep stage N3 for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
REM (rapid eye movement) latency time | 56 days
  Changes from baseline in REM (rapid eye movement) latency time for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Minimum overnight oxygen saturation index | 56 days
  Changes from baseline in minimum overnight oxygen saturation index for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Oxygen desaturation index | 56 days
  Changes from baseline in oxygen desaturation index for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Sleep related quality of life questionnaire (FOSQ) | 56 days
  Changes from baseline in the sleep related quality of life questionnaire (FOSQ - functional outcome of sleep questionnaire) for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Epworth sleepiness scale | 56 days
  Changes from baseline in patient's perception of daytime sleepiness as measured by the Epworth sleepiness scale for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Daytime sleep latency | 56 days
  Changes from baseline in daytime sleep latency time for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo
Safety of adalimumab | 56 weeks
  Evaluate the safety of adalimumab in patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Body surface area (BSA) | 56 days
  Tertiary - Changes from baseline in Body Surface Area (BSA) for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Physician's Global Assessment (PGA) | 56 days
  Tertiary - Changes from baseline in Physician's Global Assessment (PGA) for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Psoriatic Area and Severity Index (PASI) | 56 days
  Tertiary - Changes from baseline in Psoriatic Area and Severity Index (PASI) for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
PASI 75 (75% reduction in Psoriatic Area and Severity Index) | 56 days
  Tertiary - Proportion of patients who achieve PASI 75 (75% reduction in Psoriatic Area and Severity Index) at Day 56 for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Proportion with PGA (Physician's Global Assessment) of 0 or 1 | 56 days
  Tertiary - Proportion of patients who achieve a PGA (Physician's Global Assessment) of 0 or 1 at Day 56 for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.
Time to sleep induction | 56 days
  Changes from baseline in time to sleep induction for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo
Time spent in sleep stages N2 | 56 days
  Changes from baseline in time spent in sleep stages N2 for patients with psoriasis randomized to adalimumab as compared to patients randomized to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, FRCPC, Principal Investigator — Innovaderm Research Inc.
Locations (1):
- Innovaderm Research Inc., Montreal, Quebec, Canada